CLINICAL TRIAL: NCT03406156
Title: A Phase 3b Study in Previously Untreated Chronic Lymphocytic Leukemia (CLL) Subjects, Excluding Those With the 17p Deletion, to Evaluate Debulking Regimens Prior to Initiating Venetoclax Combination Therapy
Brief Title: A Study in Previously Untreated Chronic Lymphocytic Leukemia (CLL) Subjects, Excluding Those With the 17p Deletion, to Evaluate Debulking Regimens Prior to Initiating Venetoclax Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-788
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Cancer; Chronic Lymphocytic Leukemia; 17p Deletion; Debulking; Obinutuzumab; Bendamustine; Tumor lysis syndrome; Venetoclax; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Chromosome 17 deletion; Tumor Lysis Syndrome | interventions — obinutuzumab; Bendamustine Hydrochloride; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obinutuzumab (Experimental): Obinutuzumab (100 mg on Day 1 of Cycle 1, 900 mg on Day 2 of Cycle 1, and 1000 mg on Days 8 and 15 of Cycle 1 and Day 1 of Cycle 2; for Cycles 3 - 6 (1000 mg on Day 1) only as needed for participants to achieve low tumor burden) was administered via intravenous infusion during the debulking regimen.
  After debulking, obinutuzumab (1000 mg) was administered via intravenous infusion on Day 1 of one 5-week and four 4-week cycles during the obinutuzumab/venetoclax combination part of the regimen. Venetoclax was administered according to a weekly ramp-up schedule over 5 weeks to the recommended daily dose of 400 mg.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax
- Obinutuzumab/bendamustine (Experimental): Obinutuzumab (100 mg on Day 1 of Cycle 1, 900 mg on Day 2 of Cycle 1, and 1000 mg on Days 8 and 15 of Cycle 1 and Day 1 of Cycle 2; for Cycles 3 - 6 (1000 mg on Day 1) only as needed for participants to achieve low tumor burden) was administered via intravenous infusion during the debulking regimen. Bendamustine (90 mg/m^2 ) was to be administered to those with nodes or nodal mass > 10 cm, or with del(11q) and > 5 cm nodes, or at the discretion of the investigator as above, via intravenous infusion over 10 minutes on Days 1 and 2 (or Days 2 and 3 at the discretion of the investigator during Cycle 1) of each 28-day cycle for up to 6 cycles during the debulking regimen.
  After debulking, obinutuzumab (1000 mg) was administered via intravenous infusion on Day 1 of one 5-week and four 4-week cycles during the obinutuzumab/venetoclax combination part of the regimen. Venetoclax was administered according to a weekly ramp-up schedule over 5 weeks to the recommended daily dose of 400 mg.
  Interventions: Drug: Obinutuzumab; Drug: Bendamustine; Drug: Venetoclax

INTERVENTIONS:
Drug: Obinutuzumab — Administered via intravenous infusion
  Other Names: Gazyva
Drug: Bendamustine — Administered via intravenous infusion
  Other Names: Bendeka
  Arms: Obinutuzumab/bendamustine
Drug: Venetoclax — The venetoclax dose was administered according to a weekly ramp-up schedule over 5 weeks to the recommended daily dose of 400 mg. Venetoclax was continued for a total duration of up to 53 weeks, including the 5-week ramp-up schedule. Participants were instructed to take venetoclax tablets with a meal and water at approximately the same time each day. Venetoclax tablets were to be swallowed whole and not chewed, crushed, or broken prior to swallowing.
  Other Names: Venclexta; ABT-199; GDC-0199

SUMMARY:
This is a multi-cohort, open-label study in previously untreated participants with chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL), excluding those with the 17p deletion, to evaluate a debulking strategy that would enable all participants to receive subsequent venetoclax as outpatients, with lower risk of tumor lysis syndrome.

DETAILED DESCRIPTION:
Safety and efficacy data through 13 October 2021 are included in the interim analysis, which was conducted after all participants completed the post-treatment Week 65 visit or discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Adequate hematology, kidney and liver function as described in the protocol
* Diagnosis of previously untreated chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) according to 2008 Modified International Workshop on Chronic Lymphocytic Leukemia National Cancer Institute-sponsored Working Group (IWCLL NCI-WG) criteria
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 - 1
* CLL/SLL requires treatment according to the IWCLL criteria
* Medium tumor burden (any lymph node [LN] 5 to < 10 cm OR absolute lymphocyte count [ALC] ≥ 25 × 10^9/L) OR High tumor burden (any LN ≥ 10 cm OR ALC ≥ 25 × 10^9/L and LN ≥ 5 cm)

Exclusion Criteria:

* Presence of 17p deletion at Screening
* Richter's syndrome (transformation of CLL/SLL to aggressive non-Hodgkin's lymphoma or Hodgkin's lymphoma)
* Prolymphocytic leukemia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- United States (15):
  - Arizona Oncology Associates, PC-HOPE /ID# 202335, Tempe, Arizona
  - Rocky Mountain Cancer Centers - Denver Midtown /ID# 202328, Denver, Colorado
  - MidAmerica Division, Inc. /ID# 201099, Kansas City, Missouri
  - Oncology Hematology Care, Inc. /ID# 202397, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center /ID# 201201, Eugene, Oregon
  - Prisma Health Cancer Inst - Eastside /ID# 202329, Greenville, South Carolina
  - Tennessee Oncology - Chattanooga /ID# 202840, Chattanooga, Tennessee
  - Tennessee Oncology-Nashville Centennial /ID# 201098, Nashville, Tennessee
  - Texas Oncology - Austin Midtown /ID# 201199, Austin, Texas
  - Texas Oncology - Beaumont /ID# 202359, Beaumont, Texas
  - Texas Oncology - Medical City Dallas /ID# 201196, Dallas, Texas
  - Texas Oncology - McAllen /ID# 202331, McAllen, Texas
  - Texas Oncology - San Antonio Medical Center /ID# 202332, San Antonio, Texas
  - Texas Oncology - Northeast Texas /ID# 201211, Tyler, Texas
  - Northwest Cancer Specialists, P.C. /ID# 201198, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Result] Flinn IW, Andorsky D, Melear J, Manda S, Anz B III, Kolibaba K, Yimer H, Burke JM, Fanning S, Courtright J, Islas-Ohlmayer M, Kambhampati S, Vizkelety T, Pesko J, Chyla B, Jiang D, Sharman JP. Debulking Before Initiation of Venetoclax Therapy in Untreated Patients with Chronic Lymphocytic Leukemia: Results from a Phase 3b Study. American Society of Hematology - 63rd Annual Meeting. 2021
- [Result] Sharman J, Andorsky D, Melear J, Manda S, Anz B III, Kolibaba K, Yimer H, Burke J, Fanning S, Courtright J, Islas-Ohlmayer M, Kambhampati S, Jiang D, Pesko D, Vizkelety T, Sharmokh S, Nielsen J, Flinn I. Phase 3b study to evaluate debulking regimens prior to initiating venetoclax therapy in untreated patients with chronic lymphocytic leukemia. Florida Society of Clinical Oncology-2020 Fall Session
- [Result] Flinn I, Andorsky D, Melear J, Manda S, Anz B III, Kolibaba K, Yimer H, Burke J, Fanning S, Courtright J, Islas-Ohlmayer M, Kambhampati S, Jiang D, Pesko D, Vizkelety T, Sharmokh S, Sharman J. Debulking Regimens Prior To Initiating Venetoclax Therapy in Untreated Patients with Chronic Lymphocytic Leukemia: Interim Results from a Phase 3b Study. American Society of Hematology - 62nd Annual Meeting. 2020
- [Result] Sharman J, Andorsky D, Melear J, Manda S, Anz B III, Kolibaba K, Yimer H, Burke J, Fanning S, Courtright J, Islas-Ohlmayer M, Kambhampati S, Jiang D, Pesko J, Vizkelety T, Sharmokh S, Nielsen J, Flinn I. Phase 3b Study to Evaluate Debulking Regimens Prior to Initiating Venetoclax Therapy in Untreated Patients with Chronic Lymphocytic Leukemia. Society of Hematologic Oncology-8th Annual Meeting. 2020
- [Result] Sharman J, Andorsky D. Melear J, Manda S, Anz B II, Kolibaba K, Yimer H, Burke J, Fanning S, Courtright J, Islas-Ohlmayer M, Kambhampati S, Jiang D, Pesko J, Vizkelety T, Sharmkokh S, Nielsen J, Flinn I. Phase 3b study to evaluate debulking regimens prior to initiating venetoclax therapy in untreated patients with chronic lymphocytic leukemia. European Hematology Association-25th Congress. 2020
- [Result] Sharman J, Andorsky D, Melear J, Manda S, Anz B III, Kolibaba K, Yimer H, Burke J, Fanning S, Courtright J, Islas-Ohlmayer M, Kambhampati S, Al Masud A, Zimmerman T, Nielsen J, Vizkelety T, Jiang D, Flinn I. Debulking eliminates need for hospitalization prior to initiating frontline venetoclax therapy in previously untreated CLL patients: a phase 3b study. American Society of Hematology - 61st Annual Meeting. 2019
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All Treated Participants: all enrolled participants who received at least one dose of any study drug
Period: Overall Study
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Started | 84 | 36
Completed | 0 | 0
Not Completed | 84 | 36
Not completed — Death | 9 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — COVID-19 infection | 1 | 0
Not completed — Non-compliance with study procedures | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other, not specified | 72 | 28

BASELINE CHARACTERISTICS:
Population: All Treated Participants: all enrolled participants who received at least one dose of any study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine | Total
Number analyzed (Participants) | 84 | 36 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.06) | 60.7 (9.07) | 63.4 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 9 | 38
  Male | 55 | 27 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76 | 34 | 110
  Black or African American | 5 | 2 | 7
  Asian | 0 | 0 | 0
  American Indian/Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
  Missing | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Low Tumor Burden Status With Induction of Obinutuzumab or Obinutuzumab Plus Bendamustine (Debulking Period)
Description: Low tumor burden is defined as absolute lymphocyte count (ALC) < 25 × 10^9 /L and all lymph nodes < 5 cm per computed tomography (CT) scans.
Time Frame: From Baseline to the end of Cycles 2, 4, and 6, up to approximately 24 weeks after initial dose of study drug
Population: Participants who completed debulking and were subsequently treated with venetoclax with available data
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 82 | 35
percentage of participants
  From Baseline to the End of Cycle 2: number analyzed (Participants) | 59 | 31
  From Baseline to the End of Cycle 2 | 81.4 | 83.9
  From Baseline to the End of Cycle 4: number analyzed (Participants) | 60 | 31
  From Baseline to the End of Cycle 4 | 88.3 | 87.1
  From Baseline to the End of Cycle 6: number analyzed (Participants) | 60 | 31
  From Baseline to the End of Cycle 6 | 95.0 | 90.3

2. Primary Outcome: Complete Remission Rate
Description: Complete remission rate is defined as the percentage of participants achieving complete remission (CR) or complete remission with incomplete marrow recovery (CRi) as their best response based on 2008 Modified International Workshop for Chronic Lymphocytic Leukemia National Cancer Institute-Working Group (IWCLL NCI-WG) criteria.
  CR required all of the following:
  * Peripheral blood lymphocytes <4000/μL
  * Absence of lymphadenopathy by physical examination and computed tomography scan
  * No hepatomegaly or splenomegaly
  * Absence of disease or constitutional symptoms (unexplained fevers >38°C, drenching night sweats, ≥10% weight loss in last 6 months)
  * Blood counts above the following:
    * Neutrophils >1500/μL
    * Platelets >100,000/μL
    * Hemoglobin >11.0 g/dL
  * Bone marrow at least normocellular for age, <30% lymphocytes
  CRi was defined as participants with CR who had persistent cytopenia unrelated to CLL but related to drug toxicity.
Time Frame: From first dose of study drug until the last participant completed Week 65 assessments (data cut-off date of 13 October 2021); overall median time on follow-up was up to 787 days
Population: All treated participants who received at least 1 dose of any study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 84 | 36
percentage of participants | 51.2 [40.0 to 62.3] | 16.7 [6.4 to 32.8]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a best response of complete remission (CR), complete remission with incomplete marrow recovery (CRi), nodular partial remission (nPR), or partial remission (PR) based on the 2008 Modified IWCLL NCI-WG criteria at any time during the study as assessed by investigator up through the completion of the 65-week disease response assessment after the start of venetoclax. Participants who did not respond were considered non-responders.
Time Frame: as for outcome 2
Population: All treated participants who received at least 1 dose of any study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 84 | 36
percentage of participants | 94.0 [86.7 to 98.0] | 88.9 [73.9 to 96.9]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the number of days from the date of first response (CR, CRi, nPR, or PR per the 2008 Modified IWCLL NCI-WG criteria) to the date of disease progression or death, whichever occurs first. All disease progression was to be included regardless whether the event occurred during or after the participant was taking any study drug (either venetoclax, obinutuzumab, or bendamustine). Duration of response was analyzed by Kaplan-Meier (K-M) methodology.
Time Frame: as for outcome 2
Population: All treated participants who received at least 1 dose of any study drug and who had a record of first response (CR, CRi, PR, or nPR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 79 | 32
months | 21.7 [11.8 to NA] — Not calculable/estimable due to low number of participants with events | NA [NA to NA] — Not calculable/estimable due to low number of participants with events

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the number of days from the date of first dose of any study drug (either venetoclax, obinutuzumab, or bendamustine) to the date of disease progression or death, whichever occurs first. All disease progression was to be included regardless whether the event occurred during or after the participant was taking any study drug. Progression-free survival was analyzed by Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: All treated participants who received at least 1 dose of any study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 84 | 36
months | 23.3 [NA to NA] — Not calculable/estimable due to low number of participants with events | NA [17.5 to NA] — Not calculable/estimable due to low number of participants with events

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the number of days from the date of first dose of any study drug (either venetoclax, obinutuzumab, or bendamustine) to date of disease progression. All disease progression was to be included regardless of whether the event occurred during or after the participant was taking any study drug.The distribution of the time to progression was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: All treated participants who received at least 1 dose of any study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 84 | 36
months | NA [NA to NA] — Not calculable/estimable due to zero participants with events | NA [NA to NA] — Not calculable/estimable due to zero participants with events

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as number of days from the date of first dose of any study drug (either venetoclax, obinutuzumab, or bendamustine) to the date of death. If a participant had not died, their data was censored at the date when they were last known to be alive prior to the cutoff date.The distribution of OS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: All treated participants who received at least 1 dose of any study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 84 | 36
months | NA [NA to NA] — Not calculable/estimable due to low number of participants with events | NA [NA to NA] — Not calculable/estimable due to low number of participants with events

8. Secondary Outcome: Undetectable Minimal Residual Disease (UMRD) Rate
Description: The level of MRD was assessed in the peripheral blood of all participants at 5 months after last dose of obinutuzumab, and at 3 months after last dose of venetoclax/end of treatment (including early study termination) to determine the rate of UMRD. Undetectable Minimal Residual Disease is defined as less than one CLL cell per 10,000 leukocytes (< 10^-4 ).
Time Frame: From first dose of study drug until the last participant completed Week 65 assessments (data cut-off date of 13 October 2021)
Population: All treated participants who received at least 1 dose of any study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Obinutuzumab/Bendamustine
Number analyzed (Participants) | 84 | 36
percentage of participants
  At Week 38: number analyzed (Participants) | 76 | 28
  At Week 38 | 100 [95.3 to 100] | 100 [87.7 to 100]
  At Week 65: number analyzed (Participants) | 67 | 21
  At Week 65 | 95.5 [87.5 to 99.1] | 100 [83.9 to 100]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment to end of study. Median time patients were followed was: 1183.0 days (Obinutuzumab Debulking); 1185.5 days (Obinutuzumab + Bendamustine Debulking); 1114.0 days (Obinutuzumab + Venetoclax Post-debulking); and 992.5 days (Venetoclax Monotherapy Post-debulking).
Groups:
- Obinutuzumab Debulking: Participants who received obinutuzumab during the debulking regimen period
- Obinutuzumab + Bendamustine Debulking: Participants who received obinutuzumab and bendamustine during the debulking regimen period
- Obinutuzumab + Venetoclax Post-debulking: Participants who received obinutuzumab and venetoclax during the post-debulking period
- Venetoclax Monotherapy Post-debulking: Participants who received venetoclax monotherapy during the post-debulking period; safety data were collected starting 30 days after the last dose of obinutuzumab
Arm/Group | Obinutuzumab Debulking | Obinutuzumab + Bendamustine Debulking | Obinutuzumab + Venetoclax Post-debulking | Venetoclax Monotherapy Post-debulking
All-Cause Mortality (participants affected / at risk) | 1/84 | 0/36 | 1/117 | 10/114
Serious Adverse Events (participants affected / at risk) | 7/84 | 3/36 | 15/117 | 13/114
Other Adverse Events (participants affected / at risk) | 82/84 | 35/36 | 105/117 | 90/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab Debulking (N=84) | Obinutuzumab + Bendamustine Debulking (N=36) | Obinutuzumab + Venetoclax Post-debulking (N=117) | Venetoclax Monotherapy Post-debulking (N=114)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
ENDOMETRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG DISPENSED TO WRONG PATIENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab Debulking (N=84) | Obinutuzumab + Bendamustine Debulking (N=36) | Obinutuzumab + Venetoclax Post-debulking (N=117) | Venetoclax Monotherapy Post-debulking (N=114)
ANAEMIA (Blood and lymphatic system disorders) | 8 (9) | 7 (9) | 2 (3) | 1 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (6) | 3 (9) | 3 (4) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 14 (31) | 13 (27) | 35 (70) | 16 (36)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 13 (18) | 7 (10) | 11 (12) | 2 (3)
PALPITATIONS (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 11 (11) | 11 (12) | 9 (10) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 17 (24) | 11 (13) | 36 (48) | 22 (30)
DYSPEPSIA (Gastrointestinal disorders) | 6 (7) | 4 (4) | 5 (6) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 36 (46) | 21 (27) | 36 (37) | 8 (8)
VOMITING (Gastrointestinal disorders) | 5 (7) | 5 (6) | 6 (9) | 5 (6)
CHEST DISCOMFORT (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
CHILLS (General disorders) | 4 (4) | 4 (4) | 1 (1) | 6 (6)
FATIGUE (General disorders) | 37 (45) | 13 (15) | 18 (18) | 13 (17)
INFLUENZA LIKE ILLNESS (General disorders) | 7 (9) | 0 (0) | 1 (1) | 1 (2)
OEDEMA PERIPHERAL (General disorders) | 4 (5) | 3 (3) | 5 (5) | 3 (3)
PAIN (General disorders) | 4 (4) | 2 (2) | 3 (3) | 2 (2)
PYREXIA (General disorders) | 10 (12) | 10 (13) | 5 (6) | 4 (4)
BRONCHITIS (Infections and infestations) | 1 (1) | 2 (3) | 4 (4) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 6 (7) | 2 (2)
SINUSITIS (Infections and infestations) | 3 (4) | 3 (4) | 5 (6) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5) | 4 (5) | 14 (14) | 5 (6)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 6 (7) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 63 (72) | 25 (30) | 3 (3) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (8) | 4 (4) | 1 (1) | 3 (3)
BLOOD CREATININE INCREASED (Investigations) | 1 (2) | 4 (4) | 4 (4) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (2) | 2 (2) | 3 (4) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 17 (30) | 5 (7) | 22 (42) | 17 (25)
PLATELET COUNT DECREASED (Investigations) | 14 (25) | 5 (7) | 9 (13) | 4 (7)
WEIGHT DECREASED (Investigations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 4 (8) | 4 (9) | 7 (13) | 5 (6)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 1 (1) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 9 (15) | 4 (4) | 3 (9) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 1 (2) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 2 (2) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 4 (5) | 8 (8) | 1 (1) | 2 (5)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (8) | 14 (15) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 8 (9) | 5 (5)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 5 (5) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 5 (5) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 4 (4) | 2 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2) | 3 (3) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 7 (7) | 1 (2)
DIZZINESS (Nervous system disorders) | 16 (18) | 2 (2) | 5 (6) | 6 (6)
DYSGEUSIA (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 22 (25) | 9 (9) | 10 (10) | 9 (10)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
INSOMNIA (Psychiatric disorders) | 16 (19) | 3 (4) | 5 (5) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 3 (3) | 11 (14) | 10 (13)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1) | 4 (4) | 3 (3)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1) | 3 (5)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 8 (9) | 4 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 6 (6) | 5 (5)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (6) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 7 (7) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (6) | 7 (7) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (9) | 3 (3) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4) | 5 (6) | 4 (4)
HYPOTENSION (Vascular disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
PHLEBITIS (Vascular disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03406156/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT03406156/SAP_002.pdf